CLINICAL TRIAL: NCT03452475
Title: An Open-label Randomised Trial to Assess the Therapeutic Efficacy and Tolerability of Arterolane-piperaquine Plus Single Low Dose Primaquine Versus Arterolane-piperaquine Plus Mefloquine and Single Low Dose Primaquine Versus Artemether-lumefantrine Plus Single Low Dose Primaquine in the Treatment of Uncomplicated Falciparum Malaria in Children in Kenya
Brief Title: Comparison of Arterolane-piperaquine Versus Arterolane-piperaquine+Mefloquine Versus Artemether-lumefantrine in Kenyan Children
Acronym: TACTKenya
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAL17009
Record Dates: First submitted 2018-02-01; First posted 2018-03-02 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Plasmodium Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: randomised 1:1:1 to one of the three treatment arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arterolane-piperaquine (Active Comparator): Arterolane-piperaquine for 3 days
  Interventions: Drug: Arterolane-piperaquine
- Arterolane-piperaquine+mefloquine (Active Comparator): Arterolane-piperaquine + mefloquine for 3 days
  Interventions: Drug: Arterolane-piperaquine+mefloquine
- Artemether-lumefantrine (Active Comparator): Artemether-lumefantrine for 3 days
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Arterolane-piperaquine — Arterolane maleate-piperaquine phosphate tablets (37.5 mg/187.5 mg)
  Arms: Arterolane-piperaquine
Drug: Arterolane-piperaquine+mefloquine — Arterolane maleate-piperaquine phosphate tablets (37.5 mg/187.5 mg) Mefloquine tablets (250 mg)
  Arms: Arterolane-piperaquine+mefloquine
Drug: Artemether-lumefantrine — Artemether-lumefantrine tablets (20 mg/120 mg)
  Arms: Artemether-lumefantrine

SUMMARY:
This open-label randomised controlled clinical trial will compare the safety, tolerability, therapeutic efficacy and pharmacokinetics and pharmacodynamics of arterolane-piperaquine, arterolane-piperaquine plus mefloquine versus artemether-lumefantrine.in children with uncomplicated falciparum malaria in Kilifi, Kenya. This study will also provide an up to date insight on the current presence of antimalarial resistance in this site.

In addition, all children will be treated with a single low dose of primaquine, dosing is age based.

The investigators will recruit 219 patients aged 2 years to 12 years with acute uncomplicated falciparum malaria in Kilifi County Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 2 years to <13-year-old
2. Uncomplicated falciparum malaria as defined as:

   * Positive blood smear with asexual forms of P. falciparum (may be mixed with non-falciparum species)
   * Parasitaemia between 5,000-250,000 parasites/µL
   * Fever defined as tympanic temperature >37.5°C or history of fever within last 48 hours
3. Ability to take oral medication
4. Willingness and ability to comply with study protocol for study duration
5. Written informed consent given to participate in the trial

Exclusion Criteria:

1. Signs of severe/complicated malaria*
2. Any clinical reason suggesting that the child's treatment should be given immediately and not delayed during the transfer to Kilifi County Hospital in the opinion of the treating physician.
3. Acute illness other than malaria requiring urgent systemic treatment as assessed by the treating physician
4. Previous splenectomy
5. Treatment with artemisinin or ACT within the previous 7 days
6. Treatment with mefloquine in the 2 months prior to presentation
7. Known hypersensitivity or contraindication to arterolane-piperaquine, DHA-piperaquine, artemisinin, mefloquine (epilepsy, major psychiatric illness) or primaquine
8. QTc interval >450 milliseconds at point of presentation
9. Known personal or family history of cardiac conduction problems
10. Participation within another clinical trial in the previous 3 months

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 219 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
42-day PCR corrected adequate clinical and parasitological response (ACPR) by day 42 by study arm | 42 days

SECONDARY OUTCOMES:
Parasite clearance half-life | 42 days
  Parasite clearance half-life is assessed by entering the parasite counts (assessed by microscopy) in the WWARN PCE calculator
Parasite reduction rates | 24 and 48 hours
  Parasite reduction rates and ratios at 24 and 48 hours assessed by microscopy
Parasite count to fall 50% | 42 days
  Time for parasite count to fall 50% of initial parasite density
Parasite count to fall 90% | 42 days
  Time for parasite count to fall 90% of initial parasite density
Fever clearance time | 42 days
  The time taken for the tympanic temperature to fall below 37.5˚C and remain there for at least 24 hours
Incidence of clinical adverse events and serious adverse events | 42 days
Incidence of adverse events concerning markers of hepatic or renal toxicity | 42 days
  Total bilirubin, Alanine transaminase, Aspartate transaminase, Alkaline phosphatase and creatinine will be measured
Incidence of prolongation of the corrected QT interval | 42 days
  Incidence of the prolongation of the corrected QT interval above 500 ms or > 60 ms above baseline values
Prolongation of the corrected QT interval | Baseline, hour 4, hour 24, hour 28, hour 48 and hour 52
  Prolongation of the corrected QT interval compared at hour 4, hour 24, hour 28, hour 48 and hour 52 compared to baseline
Change in haematocrit | Baseline, hour 24, hour 48, hour 72, day 7, day 14, day 21, day 28, day 35 and day 42
  Change in haematocrit at hour 24, hour 48, hour 72, day 7, day 14, day 21, day 28, day 35 and day 42 according to geographical location and study arm, stratified for G6PD status
Proportion of patients that reports completing a full course of observed TACT or ACT | 42 days
  Proportion of patients that reports completing a full course of observed TACT or ACT without withdrawal of consent or exclusion from study because of drug related serious adverse event
Prevalence of Kelch13 mutations of known significance | Baseline
  Prevalence of Kelch13 mutations of known significance
Prevalence/incidence of other genetic markers of antimalarial drug resistance such as multidrug resistance gene 1 copy number and multidrug resistance gene 1 mutations | Baseline
  Prevalence/incidence of other genetic markers of antimalarial drug resistance such as multidrug resistance gene 1 copy number and multidrug resistance gene 1 mutations
Genome wide association with in vivo/in vitro sensitivity parasite phenotype | Baseline
  Genome wide association with in vivo/in vitro sensitivity parasite phenotype
A comparison of transcriptomic patterns between sensitive and resistant parasites | Baseline and 6 hours
  Transcriptomic patterns measure at baseline and at specified time points after the start of treatment comparing sensitive and resistant parasites
Proportion of patients with gametocytaemia before, during and after treatment | 42 days
  Proportion of patients with gametocytaemia before, during and after treatment
Levels of RNA transcription coding for male or female gametocytes | Baseline
  Levels of RNA transcription coding for male or female gametocytes at admission
In vitro sensitivity of P. falciparum to artemisinins and partner drugs | Baseline and day recurrent infection
Pharmacokinetic profiles and interactions (Cmax) of arterolane and partner drugs | 42 days
  Pharmacokinetic profiles and interactions (Cmax) of arterolane and partner drugs
Day 7 drug levels of partner drugs in association with treatment efficacy and treatment arm | 7 days
  Day 7 drug levels of partner drugs in association with treatment efficacy and treatment arm
Data on recent travel and current location of living | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Kilifi County Hospital, Kilifi, Kenya

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data will be entered to a database maintained by Mahidol-Oxford-Research-Unit. Individual-level anonymized data will be shared with medical regulators where appropriate. For wider stake-holder engagement and the medical community summary-level statistical analyses will be shared. Information collected or generated during this study may be anonymised for use to support new research and policies for antimalarial drug resistance. Any future research using information from this study must first be approved by a local or national expert committee to make sure that the interests of participants and their communities are protected.

REFERENCES:
- [Derived] Hamaluba M, van der Pluijm RW, Weya J, Njuguna P, Ngama M, Kalume P, Mwambingu G, Ngetsa C, Wambua J, Boga M, Mturi N, Lal AA, Khuroo A, Taylor WRJ, Goncalves S, Miotto O, Dhorda M, Mutinda B, Mukaka M, Waithira N, Hoglund RM, Imwong M, Tarning J, Day NPJ, White NJ, Bejon P, Dondorp AM. Arterolane-piperaquine-mefloquine versus arterolane-piperaquine and artemether-lumefantrine in the treatment of uncomplicated Plasmodium falciparum malaria in Kenyan children: a single-centre, open-label, randomised, non-inferiority trial. Lancet Infect Dis. 2021 Oct;21(10):1395-1406. doi: 10.1016/S1473-3099(20)30929-4. Epub 2021 Jun 7. PMID 34111412